CLINICAL TRIAL: NCT05005351
Title: "SMART-FM": Smart-Phone Based Digital Therapeutic for Management of Fibromyalgia
Acronym: SMART-FM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swing Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Swing-004
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Digital Acceptance and Commitment Therapy (ACT) (Active Comparator)
  Interventions: Device: Digital ACT
- Digital Symptom Tracker (Active Comparator)
  Interventions: Device: Digital Symptom Tracker

INTERVENTIONS:
Device: Digital ACT — Participants in Digital ACT arm complete daily ACT lessons and activities and continue their non-pharmacological and pharmacological treatment as usual.
  Arms: Digital Acceptance and Commitment Therapy (ACT)
Device: Digital Symptom Tracker — Participants in the Digital Symptom Tracker arm complete daily symptom and function tracking, have access to digital fibromyalgia and health education, and continue their non-pharmacological and pharmacological treatment as usual.
  Arms: Digital Symptom Tracker

SUMMARY:
This is a non-significant risk, multi-center, randomized, active-controlled study to compare the effectiveness of two digital therapies in the management of fibromyalgia over 12 weeks. The primary endpoint is mean change from baseline to Week 12 in the weekly revised Fibromyalgia Impact Questionnaire (FIQ-R) total score.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is 22 to 75 years of age, inclusive
2. Subject has a diagnosis of primary FM as defined by the 2016 American College of Rheumatology Preliminary Diagnostic Criteria for FM, which requires satisfaction of the following criteria:

   1. Widespread pain index (WPI) ≥7 and symptom severity (SS) scale score ≥5, OR WPI 4-6 and SS scale score ≥9;
   2. Symptoms have been present at a similar level for at least 3 months;
   3. Pain must be present in at least 4 out of 5 body regions
3. Subject with ongoing treatments should be on stable therapy for 30 days prior to screening appointment.
4. Subject is capable of reading and understanding English and has provided written informed consent to participate.

Key Exclusion Criteria:

1. Lifetime history of bipolar disorder as assessed by the MINI.
2. Current, untreated, major depressive episode and/or anxiety disorders as assessed by the MINI.
3. Subject has a BDI-II total score > 25 at either the Screening appointment or Baseline appointment.
4. The subject is at increased risk of suicide on the basis of the investigator's judgment, a response > 1 to BDI item #9, or the results of the Columbia-Suicide Severity Rating Scale ("C-SSRS") conducted at Screening or Baseline (i.e., any suicidal behavior during the preceding year or C-SSRS Type 3, 4, or 5 suicidal ideation during the preceding year).
5. Subject has any other disease or medical condition that, in the opinion of the Investigator or Sponsor, could endanger the subject, interfere with the evaluation of the study device's efficacy or safety, or compromise the subject's ability to comply with/complete the study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gendreau, MD, Study Director — Consulting Chief Medical Officer
Locations (7):
- United States (7):
  - Excell Research, Inc., Oceanside, California
  - Superior Research LLC, Sacramento, California
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Catella S, Gendreau RM, Kraus AC, Vega N, Rosenbluth MJ, Soefje S, Malhotra S, Luciano JV, McCracken LM, Williams DA, Arnold LM. Self-guided digital acceptance and commitment therapy for fibromyalgia management: results of a randomized, active-controlled, phase II pilot clinical trial. J Behav Med. 2024 Feb;47(1):27-42. doi: 10.1007/s10865-023-00429-3. Epub 2023 Jun 29. PMID 37382794
- See also: Swing Therapeutics Website — https://www.swingtherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Digital Acceptance and Commitment Therapy (ACT) Arm: Digital ACT: Participants in Digital ACT complete daily ACT lessons and activities and continue their non-pharmacological and pharmacological treatment as usual.
- Digital Symptom Tracker Arm: Digital Symptom Tracker: Participants in the Digital Symptom Tracker arm complete daily symptom and function tracking, have access to digital fibromyalgia and health education, and continue their non-pharmacological and pharmacological treatment as usual.
Period: Overall Study
Arm/Group | Digital Acceptance and Commitment Therapy (ACT) Arm | Digital Symptom Tracker Arm
Started | 39 | 28
Completed | 37 | 27
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Digital Acceptance and Commitment Therapy (ACT): Digital ACT: Participants in Digital ACT complete daily ACT lessons and activities and continue their non-pharmacological and pharmacological treatment as usual.
- Total: Total of all reporting groups
Arm/Group | Digital Acceptance and Commitment Therapy (ACT) | Digital Symptom Tracker Arm | Total
Number analyzed (Participants) | 39 | 28 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (10.5) | 53.6 (10.1) | 52.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 28 | 66
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 32 | 24 | 56
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Revised Fibromyalgia Impact Questionnaire (FIQ-R) Total Score
Description: FIQ-R total score ranges between 0-100 with a reduction in score indicating reduced fibromyalgia severity.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Digital Acceptance and Commitment Therapy (ACT) Arm | Digital Symptom Tracker Arm
Number analyzed (Participants) | 39 | 28
score on a scale | -8.7 (2.0) | -3.0 (2.4)

2. Secondary Outcome: Key Secondary Endpoint of This Clinical Trial - Rate of Patient's Global Impression of Change (PGIC) Responders at Week 12 - Any Improvement
Description: PGIC scores included are: Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Acceptance and Commitment Therapy (ACT) Arm | Digital Symptom Tracker Arm
Number analyzed (Participants) | 37 | 27
Participants | 27 | 6

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Digital Acceptance and Commitment Therapy (ACT) Arm | Digital Symptom Tracker Arm
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/28
Other Adverse Events (participants affected / at risk) | 7/39 | 3/28
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Digital Acceptance and Commitment Therapy (ACT) Arm (N=39) | Digital Symptom Tracker Arm (N=28)
COVID-19 (Infections and infestations) | 0 | 2
Sinus infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Cellulitis in Face (Infections and infestations) | 0 | 1
Post COVID-19 Vaccination Syndrome (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Broken Foot (Injury, poisoning and procedural complications) | 1 | 0
Worsening Anemia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Exacerbation of Gastroparesis (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Exacerbation of Fibromyalgia Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Left Side Rib Contusions (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-01-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT05005351/Prot_000.pdf